CLINICAL TRIAL: NCT04928053
Title: Cognition Sociale et caractéristiques Psychotiques : Approche génétique et phénomique
Brief Title: COG-PSYCHO : Social Cognition and Psychotic Characteristics: Genetic and Phenomic Approach
Acronym: COG-PSYCHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N°IDRCB 2018-A1459-46
Record Dates: First submitted 2021-02-26; First posted 2021-06-16 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Social Cognition of Schizophrenia, Bipolas or Depressed Patients
Keywords: social cognition of schizophrenia, bipolas or depressed patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phenotypic data and a blood prelevment (Experimental)
  Interventions: Genetic: ocytocine dosage and genetic analyse

INTERVENTIONS:
Genetic: ocytocine dosage and genetic analyse — All patients are assessed using 4 paradigms: Reading the Mind in the Eyes Test (RMET), Interpersonal Reactivity Index (IRI), Empathy Quotient (QE), and a modified Delay Discounting task. They have a blood prelevment

SUMMARY:
Bipolar disorder (BD), schizophrenia and depression can feature cognitive impairment, especially in social cognition (SC). According to previous studies, some genes from the oxytocin and dopamine pathways may be involved SC performance. Our endophenotype approach aimed to demonstrate that SC deficits are more severe in schizophrenia and BD or depression with psychotic symptoms (PBP) and are associated with certain Single Nucleotide Polymorphisms (SNPs) variants.

600 patients with schizophrenia, BD ou depression with and without psychotic symptoms will be recrited. Social Cognition was assessed using 4 paradigms: Reading the Mind in the Eyes Test (RMET), Interpersonal Reactivity Index (IRI), Empathy Quotient (QE), and a modified Delay Discounting task. After DNA extraction from blood or saliva sample, we used PCR amplification and real-time detection to genotype SNPs from Oxytocin pathways. he level of ocytocine will be also mesured.

DETAILED DESCRIPTION:
Schizophrenia and mood disorders represent two severe and frequent disease with heterogeneous phenotype sharing some clinical symptoms (possible presence of psychotic symptoms in mood disorders, systematic in schizophrenia) and neurocognitive impairments including social cognition. These disorders result from an interaction of several minor effect genes with various early or late environmental factors, with psychosocial or biological origin.

The association of these pathologies with dysfunctions of major neurotransmission systems has been the subject of numerous studies, but the results have often been contradictory for methodological, clinical (phenotypic heterogeneity) and finally genetic reasons. The definition of the phenotype is an essential issue in research on the genetics of mental disorders. The risk of phenotypic misclassification of subjects during genetic studies confirms the need for a better delimitation of homogeneous patient sub-populations. The development by the National Institute of Mental Health (NIMH) of clinical research criteria is essential to bring sufficient power to modern research in genetics, but also in imaging, neuroscience or behavioral sciences of mental disorders.

The aim of our work is to study a restricted phenotype of schizophrenia and mood disorders: the assessment of social cognitions. Deficits in social cognition constitute one of the subconstructs described by the NIMH and lead to functional and clinical maladjustment hindering psychosocial rehabilitation. Indeed, oxytocin is reported to be a mediator of the regulation of social cognition (including empathy and theory of mind) and emotional behaviors (Meyer-Lindenberg, 2011).

The current project involves the analysis of several social cognition tasks that measure social perception, facial recognition of affect and empathy. The objective of this work is to highlight an association between performance on the 4 social cognition paradigms and polymorphisms of the OXT and OXTR genes and in a population of subjects suffering from schizophrenia or mood disorder with or without psychotic symptoms.

The main hypothesis of this study is that these genes have an impact on social cognition in each of the populations recruited (patients with schizophrenia or patients with a mood disorder). The secondary hypothesis is to show that this impact of the genotype is more marked in patients with psychotic symptoms (suffering from mood disorders or schizophrenia) compared to patients suffering from mood disorders without psychotic symptoms (interaction mechanism).

Main objective : To show the association between variants of the OXT and OXTR genes and the deficit in social cognition observed in patients with schizophrenia or a mood disorder with or without psychotic features.

Primary endpoint : Performance on the Reading the Mind in the Eyes Test (RMET), which measures the ability to attribute emotions to others.

Secondary Objectives :

1. To show the impact of the OXT and OXTR genes on 3 other paradigms of social cognition, and in the following subgroups: schizophrenic patients, patients with mood disorders, patients with psychotic symptoms and patients without psychotic symptoms.
2. To highlight interactions between genetic variants of the OXT and OXTR genes with the main impaired cognitive and neurological capacities in schizophrenia and mood disorders (attention, executive and memory function).
3. To search for an association between traumatic life events in childhood and delusional clinical phenotype and impaired cognition in mood disorders.
4. To demonstrate that plasma oxytocin levels are decreased in patients with psychotic symptoms compared to patients without psychotic symptoms and correlated with social cognition performance in the total sample of subjects as well as in each of these subgroups.
5. To demonstrate that OXTR gene expression is reduced in patients with psychotic symptoms (schizophrenia or mood disorder with psychotic symptoms) compared to subjects without psychotic symptoms (mood disorder without psychotic symptoms), and correlated with social cognitive performance in the total sample of subjects and in each of these subgroups.

Secondary Evaluation Criteria :

1. Performance on three other tests measuring social cognitions: Delay Discouting applied to social cognitions, Interpersonal Reactivity Index and Empathy Quotient (Berthoz et al., 2008)
2. RMET test performance
3. Potentially traumatic life events (CTQ questionnaire)
4. Plasma determination of circulating oxytocin
5. mRNA expression level of the OXTR gene measured by RT-qPCR Monocentric cross-sectional study evaluating social cognition in patients suffering from schizophrenia, mood disorder with or without psychotic symptoms in search of genetic determinants involved in social cognition performance.

Patients undergo biological sampling (genotyping of variants of the OXT and OXTR genes, quantification of circulating oxytocin and quantification of OXTR transcript expression) and undergo several evaluations (RMET, Delay Discounting, Interpersonal Reactivity Index, Empathy Quotient).

Criteria for inclusion

* Major patient under 75 years of age
* Presenting the DSM-5 criteria for schizophrenia, bipolar disorder or major depressive episode.
* Capable of giving consent or under curatorship
* Benefiting from a health insurance plan Criteria for non-inclusion Pregnancy (urine test performed prior to inclusion in the program) Procedure A single three-hour face-to-face interview will be carried out at the inclusion, in an inpatient or outpatient setting. Patients will have a 30-minute social cognition assessment by the RMET, two empathy self-questionnaires: IRI and QE, and a computerized update time stamp.

The collection of standardized psychiatric and addictological diagnoses using the DIGS is under the responsibility of Professor DUBERTRET (Hôpital Louis Mourier) in order to define the groups of subjects. There is no follow-up on a day-by-day basis; patient participation is one day.

All subjects will have a blood sample in order to perform genetic analyses including genotyping of the genes tested, quantification of OXTR mRNA expressed in peripheral venous blood (biogps) by RT-qPCR and oxytocin assay.

Number of patients 600 patients

1 (monocentric study) Duration of inclusion: 5 years Duration of participation (treatment + follow-up):1 day Total research duration 5 years

ELIGIBILITY:
"Inclusion criteria :

* - Major patient under 75 years of age
* Presenting the DSM-5 criteria for schizophrenia, bipolar disorder or major depressive episode.
* Capable of giving consent or under curatorship
* Benefiting from a health insurance plan

Exclusion criteria :

* Pregnancy (urine test performed prior to inclusion in the program)
* "

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-02-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Showing an correlation between SNPs of OXT et OXTR genes and social performence observed in patients with schizophrenia and bipolar or depressed patients with or without psychotic characteristics. | 5 years
  performence at RMET (Reading the Mind in the Eyes Test)

SECONDARY OUTCOMES:
Interpersonal Reactivity Index (IRI) | 5 years
  Impact of OXT, OXTR genes and social performence emesured with Interpersonal Reactivity Index (IRI) observed in patients with schizophrenia and bipolar or depressed patients with or without psychotic characteristics.
Empathy Quotient (QE) | 5 years
  Impact of OXT, OXTR genes and social performence emesured with Empathy Quotient (QE) observed in patients with schizophrenia and bipolar or depressed patients with or without psychotic characteristics.
modified Delay Discounting task | 5 years
  Impact of OXT, OXTR genes and social performence emesured with a modified Delay Discounting task observed in patients with schizophrenia and bipolar or depressed patients with or without psychotic characteristics.
Cognitive performence | 5 years
  correlation between SNPs of OXT et OXTR genes and general cognition scores (attention, executive and mnesisic fonction)
Potentially traumatic life events (CTQ questionnaire) | 5 years
  Association between traumatic events and psychotic characteristics and cognition scores
Plasma determination of circulating oxytocin | 5 years
  - Plasma determination of oxytocin in patients with schizophrenia and bipolar, depressed patients and those without psychotic characteristics
mRNA expression level of the OXTR gene measured by RT-qPCR | 5 years
  Expression of OXT et OXTR genes reduced and associated with social performence observed in patients with schizophrenia and bipolar or depressed patients with psychotic characteristics compared with those without

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Dubertret, Principal Investigator — APHP
Locations (1):
- Hopital Louis Mourier, Colombes, France